CLINICAL TRIAL: NCT01267448
Title: A Pilot Study of Outpatient Discharge Therapy With Saxagliptin + Metformin XR or Sulphonylurea for Recently Diagnosed Type 2 Diabetes Presenting With Severe Hyperglycemia
Brief Title: Outpatient Discharge Therapy With Saxagliptin+MetforminXR vs GlipizideXL for Type 2 Diabetes With Severe Hyperglycemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cook County Health (Other Government)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Leon Fogelfeld MD, Co-Principal Investigator, Cook County Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-10-182
Record Dates: First submitted 2010-12-27; First posted 2010-12-28 (Estimated); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Diabetes Mellitus Type 2; Hyperglycemia
Keywords: Diabetes Mellitus Type2.; Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia | interventions — Glipizide; saxagliptin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saxagliptin + Metformin XR (Active Comparator): Saxagliptin 5 mg + Metformin XR 1000 mg will be automatically titrated weekly in 2 weeks to Saxagliptin 5 mg + Metformin XR 2000 daily for a total duration of 12 weeks.
  Interventions: Drug: Saxagliptin + Metformin XR; Drug: Metformin XR
- the Control goup Glipizide XL (Active Comparator): The control group will receive Sulphonylurea (Glipizide XL 10mg orally) for a total duration of 12 weeks.
  Interventions: Drug: Glipizide XL

INTERVENTIONS:
Drug: Glipizide XL — The control group will receive Glipizide XL (10mg orally) for a total duration of 12 weeks.
  Other Names: Glucotrol XL
  Arms: the Control goup Glipizide XL
Drug: Saxagliptin + Metformin XR — The intervention group will receive Saxagliptin 5 mg daily for a total duration of 12 weeks.
  Other Names: Onglyza
  Arms: Saxagliptin + Metformin XR
Drug: Metformin XR — The intervention group will receive Metformin XR 1000 mg daily and will be automatically titrated weekly in 2 weeks to Metformin XR 2000 daily for a total duration of 12 weeks.
  Other Names: Glucophage XR
  Arms: Saxagliptin + Metformin XR

SUMMARY:
Saxagliptin + Metformin XR (S+M) will be effective in stabilizing blood glucose (BG) levels in patients with newly diagnosed type 2 diabetes (T2DM) with severe hyperglycemia (BG levels 300 to 450 mg/dl) and glucose toxicity and with no criteria for inpatient admission or occurrence of severe hypoglycemia compared to glipizide XL.

The study may provide preliminary evidence to support the role of S+M as a bridging, stabilizing and safe therapy in patients with severe hyperglycemia

DETAILED DESCRIPTION:
There is very little information regarding diabetes discharge regimens for patients with recently diagnosed diabetes (<1 year duration) who present with severe hyperglycemia (blood glucose 300-450 mg/dl) to the ED or other clinical settings and who do not need to be admitted.

A combination of Saxagliptin+Metformin XR, could be a potential drug combination to be tested as an initial treatment in these circumstances compared to Glipizide XL which was shown to be effective in our previous study. We expect Saxagliptin to improve beta cell function and decrease glucagon levels as was shown for the DPP-IV class medications and in turn improve blood glucose levels, while Metformin XR may reduce insulin resistance and hepatic glucose output. Such discharge therapy may help to prevent deterioration into acute metabolic complications (DKA or hyperosmolar states) and avoid hospitalization. A high proportion of patients may achieve glycemic targets without significant hypoglycemia as measured by self glucose monitoring and objectively by continuous glucose monitoring system (CGMS). Such an easy regimen may safely bridge the time gap until patients will be seen by their providers.

ELIGIBILITY:
Inclusion Criteria:

1. Target Population

   1. Subjects recently diagnosed with T2DM (less than 1 year duration) who are either drug naïve or who had not taken oral anti-diabetic agents or insulin for more than 2 weeks.
   2. FBG and or RBG > 300mg/dl and < 450mg/dl
2. Age and Sex

   1. Men and women aged 18 to 75 years of age.
   2. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 4 weeks after the last dose of study drug to minimize the risk of pregnancy.

WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours before the start of the investigational product.

Exclusion Criteria:

1. Sex and Reproductive Status

   1. WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 4 weeks after the last dose of study drug.
   2. Women who are pregnant or breastfeeding.
   3. Women with a positive pregnancy test.
   4. Sexually active fertile men not using effective birth control if their partners are WOCBP.
2. Target Disease Exceptions

   1. Type 2 diabetes with weight less than 120 pounds
   2. Type 1 diabetes
   3. History of diabetic ketoacidosis or hyperosmolar nonketotic coma
3. Medical History and Concurrent Diseases

   1. Age >75 years
   2. History of congestive heart failure
   3. Evidence of an impaired sensorium and/or dementia
   4. Current history of alcohol or substance abuse
   5. Patients with any acute or active chronic medical illness
4. Physical and Laboratory Test Findings

   1. FBG and /or RGB < 300 mg/dl or >450 mg/dl
   2. Unstable vitals signs (temperature >101 degrees Fahrenheit, systolic blood pressure <90 or >180 mmhg, diastolic blood pressure <60 or >110 mmhg, heart rate <60 or >120 beats/minute)
   3. Electrolyte imbalances (serum bicarbonate level <20 mEq/L, serum sodium <125 or >150 mEq/L, serum potassium <3.5 or >5.5 mEq/L), serum creatinine more than 1.5 in males and 1.4 in females, creatinine clearance less than 60ml/min, liver enzymes 3 times above upper limit of normal range.
   4. HbA1c > 12% (based on our previous study (4) patients with HbA1c of >12 had a high rate of non-responders)
   5. Liver enzymes 3 times above upper limit of normal range.
   6. Allergies and Adverse Drug Reactions -Subjects with a history of any serious hypersensitivity reaction to saxagliptin, glipizide or metformin XR.
5. Prohibited Treatments and/or Therapies

   a)Treatment with systemic cytochrome P450 3A4 (CYP 3A4) inhibitors.
6. Other Exclusion Criteria

   1. Prisoners or subjects who are involuntarily incarcerated.
   2. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-09-09 (Actual); Primary Completion 2015-07-25 (Actual); Study Completion 2015-07-25 (Actual)

PRIMARY OUTCOMES:
The proportion of responders in each arm. Responder: FBG 70-300 and/or PPBG <400 mg/dl (week1-6), FBG 70-250 and/or PPBG <300 mg/dl (week 7-12) and without metabolic exclusion criteria, repeat ED visits, hospitalization or significant hypoglycemia. | 12 weeks
  Non-responder:1 FBG >300 and/or PPBG >400 mg/dl (week 1-6) and FBG >250 and/or PPBG >300 mg/dl in 4 consecutive readings or more (week 7-12).
  2. A single confirmed BG of >450 mg/dl. 3. Significant hypoglycemia: Single episode of hypoglycemia with BG < 50 mg/dl or 2 episodes of BG between 50 and 70 mg/dl within 7 days or any episode of symptomatic hypoglycemia.
  4. Persistently positive large ketones in urine and/or electrolyte imbalances. 5. Revisit to ED or admission to hospital because of hypoglycemia or uncontrolled hyperglycemia.

SECONDARY OUTCOMES:
Proportion of patients achieving FBG goal of 70-130 mg/dl at 12 weeks in the 2 treatment arms | 12 weeks
  The rate of decline in BG values (mg/dl) in the two groups over the period of twelve weeks will be analyzed using a mixed model (with random intercept) as a sensitivity analysis.
  The Kaplan-Meier (KM) curves, area under the curve,t-test and chi-square analysis will be used for analysis.
Percentage of patients with symptomatic hypoglycemia | 12 weeks
  Hypoglycemia and hospitalization rates will be compared between the 2 groups using either chi-square or Fisher exact test will be used. Binary logistic regression will be used to further analysis to identify predictors of hypoglycemia.
To measure percentage compliance with medication in the two treatment arms. | 12 weeks
  Medication compliance will be assessed by pill counting. Each patient will assigned a percentage compliance and the study groups will be compared using independent two sample t-test.
The number of fold increase in beta cell function in the 2 arms. | 12 weeks
  The early insulin response (EIR) will be calculated as the ratio of insulin to glucose response at 0 and 30 minutes (ΔI30pmol/l/ΔG30mmol/l,). The homeostasis model assessment to assess basal insulin secretion (HOMA-β cell) and insulin resistance (HOMA-IR) will be calculated. The beta cell response to OGTT will be calculated as area under the curve for glucose and insulin at 0, 30 and 60 minutes using the trapezoid rule.

CONTACTS AND LOCATIONS:
Overall Officials: Ambika Babu, MD,MS, Principal Investigator — John H Stroger Hospital of Cook County
Locations (1):
- John Stroger Hospital of Cook County, Chicago, Illinois, United States